CLINICAL TRIAL: NCT02243969
Title: Effects of Alpha-linolenic Acid on 24h-ambulatory Mean Arterial Pressure in Untreated High-normal and Stage I Hypertensive Subjects
Brief Title: Alpha-linolenic Acid and Blood Pressure
Acronym: VASALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MEC 13-3-064
Record Dates: First submitted 2014-05-19; First posted 2014-09-18 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension; Lipid Metabolism Disorders
Keywords: n-3 polyunsaturated fatty acids; Alpha-linolenic acid; Blood pressure; Vascular function
MeSH Terms: conditions — Hypertension; Lipid Metabolism Disorders | interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- flaxseed oil (rich in α-linolenic acid ) (Experimental)
  Interventions: Dietary Supplement: Flaxseed oil
- high oleic sunflower oil (Placebo Comparator)
  Interventions: Dietary Supplement: high oleic sunflower oil (HOSF)

INTERVENTIONS:
Dietary Supplement: Flaxseed oil — The flaxseed oil will be provided in vials containing 5 g of oil, and should be taken for twelve weeks during the experimental period twice a day
  Arms: flaxseed oil (rich in α-linolenic acid )
Dietary Supplement: high oleic sunflower oil (HOSF) — The HOSF will be provided in vials containing 5 g of oil, and should be taken for twelve weeks during the experimental period twice a day
  Arms: high oleic sunflower oil

SUMMARY:
Rationale: Increased intakes of n-3 long chain polyunsaturated fatty acids eicosapentanoic acid (EPA) and docosahexaenoic acid (DHA), mainly found in fatty fish, are recommended for the prevention of coronary heart disease. Alpha-linolenic acid (ALA, C18:3n-3) is the most common vegetable-oil based n-3 fatty acid. Evidence exists that ALA supplementation can also have a protective effect on the development on cardiovascular disease, but may exert its cardio protective effects through different routes. The benefit may (partly) be due to blood pressure lowering. However, evidence for beneficial effects of ALA on blood pressure is conflicting. Therefore, we propose to investigate the effect of flaxseed oil, high in ALA, using a study powered on 24-hour blood pressure, in a population with high normal blood pressure and mild hypertension.

Objective: To study the effects of flaxseed oil, rich in ALA on 24h-ambulatory mean arterial pressure (MAP) in men and women with high-normal blood pressure and mild hypertension compared to high oleic sunflower oil, poor in ALA.

Study design: Using a double blind randomized, placebo-controlled parallel design, subjects will receive at random daily 10 g of flaxseed oil or a high-oleic acid sunflower oil (HOSF) as control for twelve weeks, with a run-in period of 14 days in advance.

Study population: 72 men and women, aged 40-70 years, with untreated high-normal blood pressure and stage I hypertension and a body mass index between 25 and 35 kg/m2 will participate in the run-in and intervention period. It is estimated that 144 subject have to be screened to find 72 subjects that will enter the run-in period.

Intervention: During the run-in period, subjects will receive daily 10 g of palm super olein oil. During the intervention period subjects receive either 10 g of HOSF or flaxseed oil. All oils are provided in bottles of 5 g, one will be consumed at breakfast or lunch and one at dinner.

Main study parameters/endpoints: The main study parameter is the change in 24h-ambulatory mean arterial pressure (MAP)

ELIGIBILITY:
Inclusion Criteria:

* Quetelet-index between 25-35 kg/m2
* High-normal blood pressure defined as systolic blood pressure between 130-139 mmHg and/or diastolic blood pressure between 85-89 mmHg. Or stage I hypertension defined as systolic blood pressure between 140-159 mmHg and/or diastolic blood pressure between 90-99 mmHg.
* Mean serum total cholesterol/HDL cholesterol ratio < 8
* Mean serum triacylglycerol < 4.5 mmol/L
* Mean plasma glucose < 7.0 mmol/L

Exclusion Criteria:

* Unstable body weight (weight gain or loss >2 kg in the past 3 months)
* Use of antihypertensive or anticoagulant medication
* Indication for treatment with medication according to the Standard for cardiovascular risk management of the Dutch general practitioners community (NHG)
* Usage of non-steroidal anti-inflammatory drugs (such as aspirin, ibuprofen, naproxen) and not able or willing to stop taking them from at least 4 weeks prior to the study
* Use of medication or a diet known to affect serum lipid or glucose metabolism
* Women with expected changes in the use of oral contraceptives or estrogen replacement therapy during the study period
* Women lactating, pregnant or intend to become pregnant during study
* Active cardiovascular disease like congestive heart failure or recent (<6 months) event (acute myocardial infarction, cerebro vascular accident)
* Severe medical conditions that might interfere with the study such as diabetes mellitus, epilepsy, asthma, chronic obstructive pulmonary disease, inflammatory bowel diseases and rheumatoid arthritis
* Smoking or recently quit smoking (<1 years)
* Abuse of drugs
* More than 21 alcohol consumptions per week for men and 14 consumptions for women
* Reported intense sporting activities > 10 h/w
* Not possible or difficult to venipuncture as evidenced during the screening visits
* Use of an investigational product within the previous 30 days
* Not willing to stop the consumption of vitamin supplements, fish oil capsules or products rich in plant stanol or sterol esters 3 weeks before the start of the study
* Not willing to give up being a blood donor (or having donated blood) from 8 weeks before the start of the study and during the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
24h-ambulatory mean arterial pressure (MAP) | Baseline and end of intervention period (week 2 and 14)
  Ambulatory blood pressure measurements will be performed using an automated blood pressure device with 15-minute intervals during the day and 30-minute intervals during the night.

SECONDARY OUTCOMES:
Postprandial flow mediated dilatation (FMD) | End of intervention period (week 14)
  The brachial artery FMD will be measured in a subset (n=20 per group) of the study population. FMD will be measured before and 2 hours after a fat load.
Night, day and early morning 24h-ambulatory MAP, SBP and DBP | Baseline and end of intervention (week 2 and 14)
  Ambulatory blood pressure measurements will be performed using an automated blood pressure device with 15-minute intervals during the day and 30-minute intervals during the night.
Systolic, diastolic and MAP office blood pressure | Measured every visit (week 1,2,8,14)
  Each visit blood pressure will be measured in four-fold with 1-minute interval (the first measurement will be discarded and the last three measurement will be averaged) using a calibrated device.
The fatty-acid profile of plasma phospholipids | Baseline and end of intervention period (week 2 and 14)
  measured in fasting plasma samples

OTHER OUTCOMES:
Pulse wave velocity (PWV) | Baseline and end of intervention period (week 2 and 14)
  PWV will be determined by extending data from standard brachial artery blood pressure measurements
Retinal microvasculature | Baseline and end of intervention period (week 2 and 14)
  Measured as AV-ratio and vessel diameter from digitized analogue fundus photographs
Fasting and postprandial lipid and glucose metabolism | Every visit (week 1,2,8,14) Postprandial in subset of n=20 per group
  Postprandial glucose at time point 15,30,45,60,90,120,180,240 minutes Postprandial lipids at time point 60, 120, 180, 240 minutes
Fasting and postprandial serum biomarkers for low-grade systemic inflammation (hsCRP, IL-6) and endothelial function (sICAM-1, VCAM-1, MCP-1 and sE-Selectin) | Every visit (week 1,2,8,14) Postprandial in subset of n=20 per group at time point 60, 120, 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ronald P Mensink, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands